CLINICAL TRIAL: NCT05406908
Title: Immunogenicity and Reactogenicity of Fractionated-dose Intradermal vs Standard Intramuscular Tozinameran as the Fourth Coronavirus Disease 2019 (COVID-19) Vaccine Dose in Patients With Immune-mediated Dermatologic Diseases: a Single-blinded Randomised-controlled Parallel-grouped Non-inferiority Trial
Brief Title: Intradermal Tozinameran for Patients With Immune-mediated Dermatologic Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chutima Seree-aphinan, Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MURA2022/238; TCTR20220524004 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Bullous Dermatoses; Psoriasis; COVID-19 Vaccines
Keywords: COVID-19 Vaccine; immunogenicity; autoimmune bullous diseases; psoriasis
MeSH Terms: conditions — Skin Diseases, Vesiculobullous; Psoriasis | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fractionated-dose intradermal tozinameran (Experimental): 10 micrograms (0.1 mL) of tozinameran administered intradermally to the deltoid area of the non-dominant arm with a sterile 30-gauge needle.
  Interventions: Biological: tozinameran
- standard intramuscular tozinameran (Active Comparator): 30 micrograms (0.3 mL) of tozinameran administered intramuscularly to the deltoid area of the non-dominant arm with a sterile 25-gauge needle.
  Interventions: Biological: tozinameran

INTERVENTIONS:
Biological: tozinameran — Pfizer-BioNTech COVID-19 vaccine (Trade name: Comirnaty)

SUMMARY:
This is a randomised controlled trial conducted to prove that the immunological performance of intradermal tozinameran (i.e., Pfizer-BioNTech COVID-19 vaccine) is no worse than the standard intramuscular route in patients with immune-mediated dermatologic diseases. The side effects profile and disease activity post-vaccination will also be assessed.

DETAILED DESCRIPTION:
The standard intramuscular tozinameran is widely used as a COVID-19 vaccine booster dose, although the fractionated-dose intradermal route of the vaccine has emerged as a dose-sparing and cost-effective alternative. However, before implementing the intradermal vaccine in patients with immune-mediated dermatologic diseases, its immunogenicity should be confirmed, as many of them use long-term immunosuppressive medications, which may alter their immune responses to the vaccine. This prospective open-labelled single-blinded randomised-controlled parallel-grouped non-inferiority trial aims to determine non-inferiority in the immunogenicity of fractionated-dose intradermal tozinameran in comparison with the standard intramuscular tozinameran as the fourth COVID-19 vaccine dose in patients with immune-mediated dermatologic diseases and compare vaccine-related adverse effects between the two.

ELIGIBILITY:
Inclusion Criteria:

1. Aged equal to or more than 18 years
2. Diagnosed with psoriasis or autoimmune bullous diseases
3. Completed two-doses of the primary vaccine series and the third booster dose lasted for more than three months
4. Agree to receive the fourth COVID-19 vaccine dose as tozinameran

Exclusion Criteria:

1. History of previous COVID-19 infection
2. Positive result of COVID-19 rapid antigen test (tested upon recruitment prior to vaccination)
3. Uncontrolled disease activity
4. Non-dermatologic immune-mediated diseases
5. Congenital or acquired immunodeficiency syndrome
6. Cancer
7. Pregnant women
8. Allergy to components of tozinameran
9. Inability to give written informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of humoral immunity at Week 4 | Week 4
  Anti-Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) S1 Receptor-binding domain (RBD) Immunoglobulin G (IgG)
Change from baseline level of cellular immunity at Week 12 | Week 12
  Interferon-gamma level from SARS-CoV-2 interferon-gamma release assay (IGRA)

SECONDARY OUTCOMES:
The difference in the level of SARS-CoV-2 specific humoral immunity between 4- and 12- weeks post-vaccination | Week 4, 12
  Anti-SARS-CoV-2 S1 RBD IgG
The difference in the level of SARS-CoV-2 specific humoral immunity between 12- and 24- weeks post-vaccination | Week 12, 24
  Anti-SARS-CoV-2 S1 RBD IgG
The difference in the level of SARS-CoV-2 specific cellular immunity between 12- and 24 weeks post-vaccination | Week 12,24
  IGRA-derived interferon-gamma level
Vaccine-related adverse reactions | Week 0,1,2,3,4,8,12,24
  The percentages of participants who have local or systemic vaccine-related adverse reactions
The changes in the disease activity of psoriasis patients | Week 0,1,2,3,4,8,12,24
  Psoriasis Area Severity Index (PASI)
The changes in the disease activity of autoimmune bullous disease patients | Week 0,1,2,3,4,8,12,24
  Autoimmune Bullous Skin Disorder Intensity Score (ABSIS)
The changes in the disease activity of pemphigus patients | Week 0,1,2,3,4,8,12,24
  Pemphigus Disease Area Index (PDAI)
The changes in the disease activity of bullous pemphigoid patients | Week 0,1,2,3,4,8,12,24
  Bullous Pemphigoid Disease Area Index (BPDAI)
Disease control | Week 4,12,24
  The percentages of participants who required an adjustment of systemic treatment for disease control
COVID-19 | Any time points during the study period (i.e., up to Week 24)
  The percentages of participants who are diagnosed with COVID-19 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Chutima Seree-aphinan, MD, Principal Investigator — Division of Dermatology, Department of Internal Medicine, Faculty of Medicine Ramathibodi Hospital
Locations (1):
- Dermatology outpatient clinic, Somdech Phra Debaratana Medical Center, Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and study protocol are available from the principle investigators.
Supporting Information: Study Protocol, SAP
Time Frame: available without end date
Access Criteria: upon reasonable requests made via email.